CLINICAL TRIAL: NCT00520741
Title: A Historical-controlled, Multicenter, Double-blind, Randomized Trial to Assess the Efficacy and Safety of Conversion to Lacosamide 400 mg/Day Monotherapy in Subjects With Partial-onset Seizures
Brief Title: Trial to Demonstrate the Efficacy and Safety of Conversion to Lacosamide Monotherapy for Partial-onset Seizures
Acronym: ALEX-MT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0902; 2007-005439-27 (EudraCT Number); NCT01058954 (obsolete NCT alias)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Partial Onset Seizures; Lacosamide; Monotherapy; Vimpat
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lacosamide 400 mg/day (Experimental): Lacosamide 400 mg/day
  Interventions: Drug: Lacosamide
- Lacosamide 300 mg/day (Active Comparator): Lacosamide 300 mg/day
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — 50 mg and 100 mg tablets provided for 200 mg twice daily dosing for up to 20 weeks.
  Other Names: Vimpat
  Arms: Lacosamide 400 mg/day
Drug: Lacosamide — 50 mg and 100 mg tablets provided for 150 mg twice daily dosing for up to 20 weeks.
  Other Names: Vimpat
  Arms: Lacosamide 300 mg/day

SUMMARY:
The objective of this historical-controlled trial is to demonstrate the efficacy and safety of conversion to Lacosamide monotherapy in subjects with Partial-onset Seizures who are withdrawn from 1 to 2 marketed antiepileptic drugs.

DETAILED DESCRIPTION:
Sudden unexplained death in epilepsy have been reported in epilepsy patients. A causal relationship with the administration of antiepileptic drugs has not been established. The most important known risk factor for sudden unexplained death in epilepsy (SUDEP) is the occurrence and frequency of generalized tonic-clonic seizures (GTCS). Twenty-seven patients with only GTCS were enrolled in the conversion to monotherapy study. In this study, two patients with only GTCS had SUDEP. Due to the potential increased risk of SUDEP in patients with only GTCS in a trial setting, the 1 remaining patient with only GTCS was withdrawn from this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of Epilepsy with Simple Partial Seizures (motor component) and or Complex Partial Seizures (with or without secondary generalization)
* Must be experiencing 2 to 40 seizures per 28-day period
* Stable dose of 1 or 2 marketed antiepileptic drugs
* Second Antiepileptic Drug (AED) must be less than or equal to 50 % of the minimum recommended maintenance dose per USA product label at screening

Exclusion Criteria:

* Subject has a history of primary generalized or unclassified seizures
* Seizure disorder primarily characterized by isolated auras
* History of status epilepticus
* Seizures that are uncountable due to clustering
* Has greater than 5 seizures/day
* Subjects taking Benzodiazepines, Phenobarbital or Primidone
* Subject has Vagus Nerve Stimulation (VNS)
* Significant medical or psychiatric condition
* History of alcohol or drug abuse
* History of Ethosuximide use, Felbamate use after 1994 or Vigabatrin use after 1997

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (158):
- United States (108):
  - 48, Alabaster, Alabama
  - 10, Birmingham, Alabama
  - 18, Huntsville, Alabama
  - 42, Northport, Alabama
  - 14, Phoenix, Arizona
  - 151, Phoenix, Arizona
  - 9, Phoenix, Arizona
  - 150, Sun City, Arizona
  - 103, Tucson, Arizona
  - 102, Jonesboro, Arkansas
  - 7, Little Rock, Arkansas
  - 86, Little Rock, Arkansas
  - 120, La Habra, California
  - 156, Loma Linda, California
  - 59, Los Angeles, California
  - 76, Los Angeles, California
  - 45, Newport Beach, California
  - 21, Santa Monica, California
  - 107, Torrance, California
  - 60, Aurora, Colorado
  - 25, Fairfield, Connecticut
  - 133, Dover, Delaware
  - 37, Washington D.C., District of Columbia
  - 94, Doral, Florida
  - 108, Gainesville, Florida
  - 130, Gulf Breeze, Florida
  - 55, Maitland, Florida
  - 123, Miami, Florida
  - 132, Miami, Florida
  - 77, Orlando, Florida
  - 49, Panama City, Florida
  - 109, Pinellas Park, Florida
  - 129, Port Charlotte, Florida
  - 50, Sarasota, Florida
  - 81, Sarasota, Florida
  - 4, Tallahassee, Florida
  - 163, Tampa, Florida
  - 79, Atlanta, Georgia
  - 72, Canton, Georgia
  - 40, Savannah, Georgia
  - 58, Boise, Idaho
  - 131, Hines, Illinois
  - 146, Peoria, Illinois
  - 11, Springfield, Illinois
  - 78, Indianapolis, Indiana
  - 73, Ames, Iowa
  - 124, Manhattan, Kansas
  - 160, Wichita, Kansas
  - 23, Wichita, Kansas
  - 119, Lexington, Kentucky
  - 164, Lexington, Kentucky
  - 62, Louisville, Kentucky
  - 29, Scarborough, Maine
  - 20, Baltimore, Maryland
  - 34, Baltimore, Maryland
  - 19, Bethesda, Maryland
  - 65, Pikesville, Maryland
  - 137, Waldorf, Maryland
  - 41, Detroit, Michigan
  - 30, Golden Valley, Minnesota
  - 71, Hattiesburg, Mississippi
  - 31, Chesterfield, Missouri
  - 105, Columbia, Missouri
  - 66, St Louis, Missouri
  - 174, Omaha, Nebraska
  - 17, Lebanon, New Hampshire
  - 43, Edison, New Jersey
  - 67, Voorhees Township, New Jersey
  - 36, Albany, New York
  - 83, Buffalo, New York
  - 69, Cedarhurst, New York
  - 154, Mineola, New York
  - 122, New York, New York
  - 27, New York, New York
  - 175, Schenectady, New York
  - 3, Asheville, North Carolina
  - 63, Durham, North Carolina
  - 152, Rocky Mount, North Carolina
  - 117, Wilmington, North Carolina
  - 47, Winston-Salem, North Carolina
  - 15, Cleveland, Ohio
  - 61, Columbus, Ohio
  - 2, Toledo, Ohio
  - 147, Oklahoma City, Oklahoma
  - 8, Medford, Oregon
  - 157, Portland, Oregon
  - 100, Greensburg, Pennsylvania
  - 32, Philadelphia, Pennsylvania
  - 26, Tarentum, Pennsylvania
  - 24, Beaufort, South Carolina
  - 114, Chattanooga, Tennessee
  - 1, Nashville, Tennessee
  - 138, Austin, Texas
  - 111, Dallas, Texas
  - 22, Dallas, Texas
  - 46, El Paso, Texas
  - 51, Houston, Texas
  - 53, Houston, Texas
  - 98, San Antonio, Texas
  - 82, Temple, Texas
  - 136, Layton, Utah
  - 161, Alexandria, Virginia
  - 16, Charlottesville, Virginia
  - 106, Richmond, Virginia
  - 125, Winchester, Virginia
  - 74, Renton, Washington
  - 80, Madison, Wisconsin
  - 28, Milwaukee, Wisconsin
- Australia (7):
  - 421, Capmerdown, New South Wales
  - 425, Chatswood, New South Wales
  - 423, Herston, Queensland
  - 422, Maroochydore, Queensland
  - 420, Adelaide, South Australia
  - 429, Clayton, Victoria
  - 427, Parkville, Victoria
- 204, Innsbruck, Austria
- Canada (7):
  - 127, Calgary, Alberta
  - 140, Halifax, Nova Scotia
  - 116, Hamilton, Ontario
  - 93, London, Ontario
  - 91, Greenfield Park, Quebec
  - 110, Montreal, Quebec
  - 113, Montreal, Quebec
- Denmark (2):
  - 223, Aarhus
  - 220, Copenhagen
- France (3):
  - 402, Bron
  - 404, Dijon
  - 405, Ramonville-Saint-Agne
- Germany (2):
  - 465, Berlin
  - 461, Mainz
- 240, Dublin, Ireland
- Italy (8):
  - 442, Bologna
  - 449, Catanzaro
  - 443, Ferrara
  - 441, Milan
  - 450, Perugia
  - 448, Pisa
  - 445, Reggio Calabria
  - 447, Torrette Di Ancona
- Poland (9):
  - 284, Częstochowa
  - 286, Gdansk
  - 282, Gdynia
  - 280, Krakow
  - 283, Lublin
  - 290, Lublin
  - 289, Szczecin
  - 281, Warsaw
  - 287, Warsaw
- 158, San Juan, Puerto Rico
- Spain (2):
  - 323, Granada
  - 324, Santa Cruz de Tenerife
- United Kingdom (7):
  - 360, Blackpool
  - 364, London
  - 369, London
  - 361, Manchester
  - 363, Middlesbrough
  - 368, Stoke-on-Trent
  - 367, Truro

REFERENCES:
- [Derived] Wechsler RT, Li G, French J, O'Brien TJ, D'Cruz O, Williams P, Goodson R, Brock M; ALEX-MT Study Group. Conversion to lacosamide monotherapy in the treatment of focal epilepsy: results from a historical-controlled, multicenter, double-blind study. Epilepsia. 2014 Jul;55(7):1088-98. doi: 10.1111/epi.12681. Epub 2014 Jun 10. PMID 24915838
- See also: FDA safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 160 sites in the United States of America (USA), Canada, Europe, and Australia.The maximum duration of a subject's trial participation is 30 weeks.
  The Participant Flow refers to the Safety Set (SS) population which consists of all patients who received at least one dose of study medication.
Pre-assignment Details: Subjects were randomized 3:1 to one of two therapeutic doses of Lacosamide, 400 mg/day or 300 mg/day, to ensure a study design comparable to the historical control.
Groups:
- Lacosamide 300 mg/Day: Lacosamide 300 mg/day
  Lacosamide : 50 mg and 100 mg tablets provided for 150 mg twice daily dosing for up to 20 weeks.
  Subjects were randomized 3:1 to one of two therapeutic doses of Lacosamide, 400 mg/day or 300 mg/day, to ensure a study design comparable to the historical control.
- Lacosamide 400 mg/Day: Lacosamide 400 mg/day
  Lacosamide : 50 mg and 100 mg tablets provided for 200 mg twice daily dosing for up to 20 weeks.
  Subjects were randomized 3:1 to one of two therapeutic doses of Lacosamide, 400 mg/day or 300 mg/day, to ensure a study design comparable to the historical control.
Period: Overall Study
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Started | 106 | 319 (One subject was randomized at 2 sites and excluded from the Safety Set.)
Completed | 69 | 194
Not Completed | 37 | 125
Not completed — Adverse Event | 16 | 56
Not completed — Lack of Efficacy | 11 | 30
Not completed — Withdrawal by Subject | 0 | 11
Not completed — Protocol Violation | 2 | 15
Not completed — Unsatisfactory compliance of subject | 4 | 3
Not completed — Lost to Follow-up | 4 | 4
Not completed — Other reasons for premature termination | 0 | 6

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set (SS) which includes the unique randomized subjects who took at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day | Total
Number analyzed (Participants) | 106 | 319 | 425
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 7 | 10
  Between 18 and 65 years | 99 | 303 | 402
  >=65 years | 4 | 9 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (14.3) | 40.4 (12.5) | 40.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 169 | 219
  Male | 56 | 150 | 206
Race/Ethnicity, Customized [Number; unit: participants]
  White | 91 | 246 | 337
  Black | 9 | 53 | 62
  Asian | 0 | 1 | 1
  Other | 6 | 19 | 25
Height [Mean (Standard Deviation); unit: centimeter] | 169.72 (10.69) | 169.01 (10.87) | 169.19 (10.82)
Weight [Mean (Standard Deviation); unit: kilogram] | 81.62 (19.53) | 82.13 (21.30) | 82.00 (20.85)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.22 (5.74) | 28.67 (6.64) | 28.56 (6.42)
Average Baseline Seizure Frequency per 28 days [Mean (Standard Deviation); unit: seizures/28 days] | 10.10 (8.82) | 10.22 (8.88) | 10.19 (8.86)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects (Using Kaplan-Meier) Who Are Identified As Meeting At Least 1 Pre-defined Exit Criteria By Day 112 Relative To The Start of Withdrawal of Background Antiepileptic Drug(s)
Description: Pre-defined exit criteria:
  1. A 2-fold or greater increase in average monthly (28-day) partial seizure frequency (motor and non-motor) compared to average monthly partial seizure frequency (motor and non-motor) during the Baseline Phase
  2. A 2-fold or greater increase in consecutive 2-day partial seizure frequency (motor and non-motor) versus the highest consecutive 2-day partial seizure frequency (motor and non-motor) that occurred during the Baseline Phase.
     Note: if the highest consecutive 2-day partial seizure frequency during the Baseline Phase is 1, a 2-day partial seizure frequency of ≥3 is required to meet this exit criterion
  3. Occurrence of a single generalized tonic-clonic seizure if none had occurred in the 6 months prior to randomization
  4. A prolongation or worsening of overall seizure duration, frequency, type or pattern considered by the investigator as serious enough to warrant trial discontinuation
  5. Status epilepticus, or new onset of serial/cluster seizures
Time Frame: 16 Weeks Maintenance Period (approximately 112 days)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS included subjects who completed the Titration Phase and started withdrawing background Anti-epileptic Drugs (AEDs) (ie, entered the Maintenance Phase and took at least 1 dose of Maintenance medication).
  The primary analysis is only conducted on the Lacosamide 400 mg/day group.
Measure: Number; unit: percentage of subjects
Groups:
- Lacosamide 300 mg/Day: Lacosamide (LCM) 300 mg/day
  Lacosamide : 50 mg and 100 mg tablets provided for 150 mg twice daily dosing for up to 20 weeks.
  Subjects were randomized 3:1 to one of two therapeutic doses of Lacosamide, 400 mg/day or 300 mg/day, to ensure a study design comparable to the historical control.
- Lacosamide 400 mg/Day: Lacosamide (LCM) 400 mg/day
  Lacosamide : 50 mg and 100 mg tablets provided for 200 mg twice daily dosing for up to 20 weeks.
  This study had a single inferential test of the primary efficacy variable for the LCM 400 mg/day treatment arm which was to be compared to an external historical control. As such, no adjustment for multiplicity was required. Additional analyses of the primary efficacy variable for the LCM 400 mg/day and LCM 300 mg/day treatment arms was for exploratory or supportive purposes only. The analysis of the LCM 300 mg/day arm is exploratory due to the 3:1 randomization ratio. Therefore the LCM 300 mg/day arm is not reported for this Outcome Measure.
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 0 | 284
percentage of subjects |  | 30.0
Statistical Analysis 1: Comparison: Lacosamide 400 mg/Day; The upper limit of the Confidence Interval for the estimate of the Lacosamide (LCM) 400 mg/day exit rate was compared with the lower bound of the 95 % prediction interval for the historical-control of 0.653; hereafter referred to as the historical-control exit rate. The LCM 400 mg/day dose group would be declared an effective conversion to monotherapy treatment if the upper 95 % confidence limit for the estimate of the exit rate was less than 0.653; Test type: Superiority or Other; Kaplan-Meier; Subjects who dropped out due to non-exit criteria reasons over the 10 % censoring maximum were to be counted as an exit; Predicted exit rate at 112 days = 0.300, 95% CI 2-sided [0.246 to 0.355]

2. Secondary Outcome: Time to First Occurrence of Any Exit Event During The Maintenance Period
Description: The time to first occurrence (days) of any exit event was estimated using Kaplan-Meier methods and was based on the time from the start of the Maintenance Phase to the earliest date a subject met an exit criterion. Subjects who discontinued during the Maintenance Phase due to non-exit criteria reasons or who completed the Maintenance Phase before 112 days and did not meet an exit criterion were censored as of the last Maintenance Phase dose date. Subjects completing 112 days in the Maintenance Phase were censored as of Day 112.
Time Frame: 16 Weeks Maintenance Period (approximately 112 days)
Population: The Analysis Population refers to a subset of the Full Analysis Set (FAS). The FAS included subjects who completed the Titration Phase and started withdrawing background Anti-epileptic Drugs (AEDs). In addition to being a member of FAS, subjects also met at least one of the exit criterion noted under the Primary Outcome Measure.
Measure: Median (Full Range); unit: days
Groups:
- Lacosamide 400 mg/Day: Lacosamide (LCM) 400 mg/day
  Lacosamide : 50 mg and 100 mg tablets provided for 200 mg twice daily dosing for up to 20 weeks.
  Subjects were randomized 3:1 to one of two therapeutic doses of Lacosamide, 400 mg/day or 300 mg/day, to ensure a study design comparable to the historical control.
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 26 | 82
days | 39 (21.2) [1 to 80] | 45.0 (24.3) [3 to 102]

3. Secondary Outcome: Percentage of Subjects (Using Kaplan-Meier) Who Are Identified as Meeting at Least 1 Pre-defined Exit Criteria by Day 112, Withdrew Due to Adverse Event (AE) or Withdrew Due to Lack of Efficacy During The Maintenance Period
Description: Subjects were classified as having an exit event if they experienced at least 1 of the following events during the Maintenance Phase as of Day 112:
  1. Met at least 1 exit criterion based on the calculations applied for the Primary Efficacy Analysis
  2. Withdrawal due to AE with onset during the Maintenance Phase
  3. Withdrew prematurely due to lack of efficacy during the Maintenance Phase
  The date the subject experienced the event was set to the earliest date the subject met an exit criterion or the date of the last Maintenance Phase dose for subjects not meeting an exit criterion but withdrawing due to an AE or lack of efficacy.
  The secondary analysis is only conducted on the Lacosamide 400 mg/day group.
Time Frame: 16 Weeks Maintenance Period (approximately 112 days)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS included subjects who completed the Titration Phase and started withdrawing background Anti-epileptic Drugs (AEDs) (eg, entered the Maintenance Phase and took at least 1 dose of Maintenance medication).
Measure: Number; unit: percentage of subjects
Groups:
- Lacosamide 400 mg/Day: Lacosamide (LCM) 400 mg/day
  Lacosamide : 50 mg and 100 mg tablets provided for 200 mg twice daily dosing for up to 20 weeks.
  This study had a single inferential test of the primary efficacy variable for the LCM 400 mg/day treatment arm which was to be compared to an external historical control. As such, no adjustment for multiplicity was required. Additional analyses of the primary efficacy variable for the LCM 400 mg/day and LCM 300mg/day treatment arms was for exploratory or supportive purposes only. The analysis of the LCM 300 mg/day arm is exploratory due to the 3 :1 randomization ratio. Therefore the LCM 300 mg/day arm is not reported for this Outcome Measure.
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 0 | 284
percentage of subjects |  | 32.3
Statistical Analysis 1: Comparison: Lacosamide 400 mg/Day; The upper limit of the Confidence Interval for the estimate of the Lacosamide (LCM) 400 mg/day exit rate was compared with the historical-control exit rate. The LCM 400 mg/day dose group would be declared an effective conversion to monotherapy treatment if the upper 95 % confidence limit for the estimate of the exit rate was less than 0.653; Test type: Superiority or Other; Kaplan-Meier; Subjects who dropped out due to non-exit criteria reasons over the 10 % censoring maximum were to be counted as an exit; predicted exit rate at 112 days = 0.323, 95% CI 2-sided [0.268 to 0.378]

4. Secondary Outcome: Duration of Monotherapy Treatment During the Monotherapy Phase of The Maintenance Period (Visit 9 - Visit 12)
Description: Days on Monotherapy Treatment were defined as the number of days during the Monotherapy Phase when the subject took Lacosamide (LCM) only (ie, the total number of days exposed to LCM during the Monotherapy Phase minus any days where a concomitant or rescue Anti-epileptic Drug (AED) was taken by the subject). The days on Monotherapy Treatment did not need to be consecutive.
Time Frame: Visit 9 - Visit 12 (approximately 10 weeks)
Population: The Analysis Population refers to a subset of the Full Analysis Set (FAS). The FAS included subjects who completed the Titration Phase and started withdrawing background Anti-epileptic Drugs (AEDs).This subset of the FAS included subjects who entered the Maintenance Phase but who never achieved Lacosamide (LCM) monotherapy.
Measure: Median (Full Range); unit: days
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 86 | 254
days | 71 (22.0) [1 to 100] | 71 (20.3) [2 to 105]

5. Secondary Outcome: Clinical Global Impression of Change (CGIC) From Baseline To Last Visit
Description: For the assessment of the Clinical Global Impression of Change (CGIC), the investigator should provide his/her assessment of the subject's clinical status, compared to Baseline, including an evaluation of seizure frequency and intensity, the occurrence of AEs, and subject's functional status. He was asked the following:Please check the number that best describes the subject's condition over the past 4 weeks compared to Baseline:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: Baseline; Last Visit (approximately 27 weeks)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 99 | 284
participants
  Very much improved | 21 | 56
  Much improved | 33 | 116
  Minimally improved | 18 | 42
  No change | 8 | 18
  Minimally worse | 6 | 16
  Much worse | 8 | 23
  Very much worse | 1 | 1
  Not done | 4 | 12

6. Secondary Outcome: Patient's Global Impression of Change (PGIC) From Baseline To Last Visit
Description: For the assessment of the Patient's Global Impression of Change, the subject should provide his/her assessment of his/her own clinical status, compared to Baseline, including an evaluation of seizure frequency and intensity, the occurrence of AEs, and subject's functional status.The subject was asked to answer the following:
  Over the past 4 weeks, how have you felt compared to before you entered this clinical trial? (Please check the number that best describes your condition.)
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: Baseline; Last Visit (approximately 27 weeks)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 99 | 284
participants
  Very much improved | 24 | 81
  Much improved | 33 | 93
  Minimally improved | 15 | 37
  No change | 10 | 15
  Minimally worse | 3 | 19
  Much worse | 7 | 22
  Very much worse | 3 | 3
  Not done | 4 | 14

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (week -8) up to the end of the study (week 22). Only Treatment-Emergent Adverse Events (TEAEs) are presented.
Description: Further detailed information about Sudden Unexplained Death in Epilepsy (SUDEP) is reported in the "Detailed Description" section.
Arm/Group | Lacosamide 300 mg/Day | Lacosamide 400 mg/Day
Serious Adverse Events (participants affected / at risk) | 4/106 | 21/319
Other Adverse Events (participants affected / at risk) | 74/106 | 215/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide 300 mg/Day (N=106) | Lacosamide 400 mg/Day (N=319)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Polytraumatism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 6 (6)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Toxic induced encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide 300 mg/Day (N=106) | Lacosamide 400 mg/Day (N=319)
Vision blurred (Eye disorders) | 6 (6) | 19 (25)
Nausea (Gastrointestinal disorders) | 13 (16) | 46 (57)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 21 (22)
Vomiting (Gastrointestinal disorders) | 2 (2) | 23 (27)
Fatigue (General disorders) | 12 (14) | 32 (37)
Nasopharyngitis (Infections and infestations) | 7 (8) | 28 (30)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 16 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (13)
Dizziness (Nervous system disorders) | 19 (26) | 86 (121)
Headache (Nervous system disorders) | 21 (32) | 45 (58)
Convulsion (Nervous system disorders) | 17 (22) | 29 (36)
Somnolence (Nervous system disorders) | 15 (19) | 29 (35)
Tremor (Nervous system disorders) | 8 (8) | 23 (23)
Cognitive disorder (Nervous system disorders) | 7 (8) | 6 (6)
Insomnia (Psychiatric disorders) | 8 (10) | 17 (17)
Anxiety (Psychiatric disorders) | 7 (8) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days